CLINICAL TRIAL: NCT04719416
Title: Effects of Guided Meditation on Patient Outlook and Symptom Management in Pediatric Oncology Patients
Brief Title: Relaxation Therapy in Pediatric Oncology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Other projects and needs of study personnel
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Santisree Tanikella, Physician Pediatrics, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1017
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Pediatric Cancer
Keywords: pediatric cancer; relaxation therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Treatment with Relaxation (Active Comparator): This subgroup comprises of patients who are currently receiving active treatment for their cancer diagnosis. They will be completing the pre-recorded relaxation audio therapy twice weekly prior to falling asleep.
  Interventions: Behavioral: Guided Meditation
- Remission with Relaxation (Active Comparator): This subgroup comprises of patients who are currently in remission for their cancer diagnosis. They will be completing the pre-recorded relaxation audio therapy twice weekly prior to falling asleep.
  Interventions: Behavioral: Guided Meditation
- Active Treatment without (No Intervention): This subgroup comprises of patients who are currently receiving active treatment for their cancer diagnosis. They will not be asked to complete any additional relaxation therapy.
- Remission without (No Intervention): This subgroup comprises of patients who are currently in remission for their cancer diagnosis. They will not be asked to complete any additional relaxation therapy.

INTERVENTIONS:
Behavioral: Guided Meditation — Approximately 10 minute recording of guided meditation focuses on muscle relaxation.
  Arms: Active Treatment with Relaxation; Remission with Relaxation

SUMMARY:
This study will look at the use of relaxation therapy in children with cancer. The study will compared patients who are current receiving treatment for their cancer and those who are currently in remission. Patients will be asked to listen to a short audio recording twice a week prior to going to bed which will walk patients through a mediation session. Surveys will be distributed through parental emails on the first of each month for each child to complete for the duration of 12 months. It is anticipated that the use of relaxation therapy will help to improve anxiety and pain levels in this population.

DETAILED DESCRIPTION:
Rationale: The utilization of complementary therapies in the management of cancer have not been extensively studied in the pediatric population. Patients in active treatment and even those in remission may experience higher levels of anxiety and medical complications compared to their counterparts. Complementary therapies such as meditation have been found to improve symptoms and decrease anxiety and pain levels in adult oncology patients.

Objective: The goal of this study is to determine the impact of relaxation breathing with body scan techniques through the utilization of media clips on pediatric oncology patients' complications, hospitalizations, anxiety levels and outlook on diagnosis and treatment management.

Methods: A randomized non-blind control trial will be conducted in order to compare a control to a therapy intervention group. The therapy will consist of a video clip approximately 5 minutes in length. The clip will walk the patient through mindfulness in breathing along with muscle relaxation of each muscle group. This therapy is to be completed three times a week prior to falling asleep. Prior to initiation of therapy a baseline questionnaire will be completed. Following initiation, a follow up survey will be distributed on a monthly basis to assess for symptom severity, number of hospitalizations and patient outlook.

Population: The study population includes patients seen at Janet Weis Children's Hospital's pediatric oncology clinic. Patients must be in the age range of 6-20 years old for the entire year of the study in order to qualify. Exclusion criteria includes patients who are actively receiving drug therapy for anxiety or depression or receiving palliative care. Patients who pass away within the year of study will be excluded.

Time Frame: Following recruitment, each patient will be enrolled for the total of a one-year time frame.

Expected Outcomes: The investigators project that the patients utilizing guided meditation will experience decreased levels of anxiety, pain and complications compared to those of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Current patient at Geisinger Foss Clinic - oncology department with a diagnosis of cancer for more than 2 months prior to the study start

Exclusion Criteria:

* Current use of any psychiatric medications including those for anxiety, depression or mood disorders
* Non-English speaking
* Patients receiving palliative care
* Patients with Langerhans' cell histiocytosis, benign teratomas and craniopharyngioma as they do not clearly constitute malignancy
* Patients with a history of cognitive developmental delay

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Improved anxiety level | Measurement will be assessed through study completion, an average of 1 year
  Anxiety level will be measured through a series of monthly surveys asking patients to rate how often they experience worry over their diagnosis, school, have difficulty paying attention, feel angry, sad or alone as never, rarely, sometimes or often.

SECONDARY OUTCOMES:
Improved sleep habits | Measurement will be assessed through study completion, an average of 1 year
  Sleep habits will be measured through a series of monthly surveys asking patients to rate how often they experience difficulty falling asleep, staying asleep and if they feel more tired than usual as yes or no.
Change in levels of pain | Measurement will be assessed through study completion, an average of 1 year
  Levels of pain will be assessed through monthly surveys asking the patient to rate their overall pain level over the past month as 1-10 with 10 being a lot of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Santisree Tanikella, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No